CLINICAL TRIAL: NCT05908435
Title: Measuring the Impact of Free Sunscreen Dispensers in Community Settings Frequented by Youth
Brief Title: Impact of Sunscreen Dispensers in Parks Visited by Teenagers
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Alan Geller, Alan Geller, RN, MPH, Harvard School of Public Health (HSPH)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: IRB22-1402
Record Dates: First submitted 2023-05-30; First posted 2023-06-18 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Skin Neoplasm; Adolescent Behavior; Sunscreening Agents
Keywords: Skin Neoplasm; Adolescent Behavior; Sunscreening Agents
MeSH Terms: conditions — Skin Neoplasms; Adolescent Behavior

STUDY DESIGN:
Who Masked: Participant
Masking Description: Teen survey participants will not know whether the park where the free sunscreen dispenser is located is an intervention or control site.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dispensers, Flyers, Enhanced Signage + a social media component delivered by teen ambassadors (Experimental): The DFS+ experimental group is designed to increase utilization of free sunscreen dispensers, applying and reapplying sunscreen, and motivating use of other forms of sun protection by teens in 8 Boston parks and 2 Maine beaches. IMPACT Melanoma will install and maintain free sunscreen dispensers at the study sites. Flyers will be posted at locations at the park/beach to inform people of the availability of free sunscreen and the location of the dispenser. 'Teen enhanced' signage will be present on the dispenser in the intervention parks/beaches. Teen ambassadors will share 3-5 posts to their social media platform over the course of 1 week encouraging sun protection practices and use of the free sunscreen dispenser (when the intervention is occurring at the study site).
  Interventions: Behavioral: Dispensers, Flyers, Enhanced Signage + a social media component delivered by teen ambassadors
- Dispensers, Flyers, Signage (No Intervention): The DFS control group includes dispensers, flyers, and standard signage at 8 Boston parks and 2 Maine beaches. IMPACT Melanoma will install and maintain free sunscreen dispensers at the study sites. Flyers will be posted at locations at the park/beach to inform people of the availability of free sunscreen and the location of the dispenser. Standard signage will be present on the dispenser in the control parks/beaches.

INTERVENTIONS:
Behavioral: Dispensers, Flyers, Enhanced Signage + a social media component delivered by teen ambassadors — The study intervention is designed to increase utilization of free sunscreen dispensers, applying and reapplying sunscreen, and motivating use of other forms of sun protection by teens. IMPACT Melanoma will install and maintain free sunscreen dispensers at the study sites. Flyers will be posted at locations at the park/beach to inform people of the availability of free sunscreen and the location of the dispenser. 'Teen enhanced' signage will be present on the dispenser in the intervention parks/beaches. Teen ambassadors will share 3-5 posts to their social media platform over the course of 1 week encouraging sun protection practices and use of the free sunscreen dispenser (when the intervention is occurring at the study site).
  Arms: Dispensers, Flyers, Enhanced Signage + a social media component delivered by teen ambassadors

SUMMARY:
This study will evaluate the use of publicly available free sunscreen dispensers at Maine beaches and Boston and Cambridge parks.

Aim 1: Determine the impact of DFS+ (dispensers, flyers, enhanced signage, + a social media component delivered by teen ambassadors) sun protection education on the use of free sunscreen dispensers by adolescents ages 12-20 compared with DFS (dispensers, flyers, standard signage).

Aim 2: Outcomes evaluation to assess the effects of the sunscreen dispensers and the sun-safety educational intervention on sun protection knowledge, attitudes, beliefs, and behaviors within the community.

Aim 3: Cost Evaluation and Cost-Effectiveness Analysis

DETAILED DESCRIPTION:
The investigators will build on the pioneering work of IMPACT Melanoma which has provided free sunscreen dispensers to a general population. This study will build on IMPACT Melanoma's ability to install, maintain, and now for the first time, target and publicize the use of dispensers for a teen population. The investigators will test scalable methods for improving the use of free sunscreen dispensers by testing DFS interventions compared with the addition of social media led by teen ambassadors. The investigators will evaluate the impact of the intervention in both parks and beaches in Boston, MA, Cambridge, MA and Maine.

ELIGIBILITY:
Inclusion Criteria:

* Being a Boston, MA, Cambridge, MA or Maine youth ages 12-20
* Able to complete a survey in English

Exclusion Criteria:

* Not a Boston, MA, Cambridge, MA or Maine youth ages 12-20
* Not able to complete a survey in English

Ages: 12 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1200 (Estimated)
Dates: Start 2023-06-03 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Dispenser utilization/Measured reduction in sunscreen levels in dispensers | In real-time, up to 1 day
  The investigators will count of the number of teens between the ages of 12 and 20 using the sunscreen dispenser in real-time at the park or beach as they are using the dispenser. This will serve as the numerator. The investigators will also conduct observations to determine an estimated number of teens who are the park on a given day. This will serve as the denominator. This count will be in real-time, counting the number of teens who we observe at the park or beach where the study is taking place.
Reported use of sunscreen from surveys completed by teens | In real-time, up to 1 day
  Survey responses about sunscreen use

SECONDARY OUTCOMES:
Sun prevention practices | In real-time, up to 1 day
  Survey responses about sun protection practices

CONTACTS AND LOCATIONS:
Overall Officials: Alan Geller, MPH, RN, Principal Investigator — Harvard School of Public Health (HSPH)
Locations (1):
- Harvard TH Chan School of Public Health, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No